CLINICAL TRIAL: NCT03267628
Title: Quadratus Lumborum Type 2 Block Versus Intrathecal Morphine for Analgesia Following Elective Caesarean Sections
Brief Title: Comparison of Intrathecal Morphine With the Quadratus Lumborum Type 2 Block for Post-operative Analgesia Following Elective Caesarean Section (QLBvITM Study)
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: We at the Sunshine Coast University Hospital are unable to cope with the extra effort/time needed to complete this trial properly.
Sponsor: Dr Willem Basson (Other)
Collaborators: Sunshine Coast Hospital and Health Service (Other)
Responsible Party: Sponsor-Investigator, Dr Willem Basson, Staff Specialist in Anaesthetics, Sunshine Coast Hospital and Health Service
Organization: Sunshine Coast Hospital and Health Service (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: HREC/17/QPCH/121
Record Dates: First submitted 2017-08-10; First posted 2017-08-30 (Actual); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Cesarean Section; Pain, Acute
Keywords: intrathecal morphine; quadratus lumborum type 2 block; cesarean section; pain
MeSH Terms: conditions — Acute Pain; Pain | interventions — Anesthesia, Local; Dental Occlusion; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: 4 groups of 25 patients each. All patients will receive a spinal and a quadratus lumborum type 2 block. The groups will have a combination of ITM / QLB or both or neither.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Saline intrathecal as well as saline in Blocks (Sham Comparator): These 25 patients will receive 0.3ml saline added to the spinal anaesthetic and 25 ml saline both sides as a QLB2.
  Interventions: Procedure: Saline intrathecal as well as saline in Blocks; Procedure: Saline intrathecal as well as local anaesthetic in Blocks
- Saline intrathecal as well as local anaesthetic in Blocks (Active Comparator): These 25 patients will receive 0.3ml saline added to the spinal anaesthetic and 25 ml local anaesthetic both sides as a QLB2.
  Interventions: Procedure: Intrathecal morphine as well as local anaesthetic in Blocks; Procedure: Saline intrathecal as well as saline in Blocks
- Intrathecal morphine as well as local anaesthetic in Blocks (Active Comparator): These 25 patients will receive 0.3ml (150mcg) morphine added to the spinal anaesthetic and 25 ml local anaesthetic both sides as a QLB2.
  Interventions: Procedure: Intrathecal morphine as well as local anaesthetic in Blocks; Procedure: Intrathecal morphine as well as saline in Block
- Intrathecal morphine as well as saline in Block (Active Comparator): These 25 patients will receive 0.3ml (150mcg) morphine added to the spinal anaesthetic and 25 ml saline both sides as a QLB2.
  Interventions: Procedure: Intrathecal morphine as well as saline in Block; Procedure: Saline intrathecal as well as local anaesthetic in Blocks

INTERVENTIONS:
Procedure: Intrathecal morphine as well as local anaesthetic in Blocks — A Quadratus lumborum type 2 block will be performed under ultrasound with 25 ml 0.375% ropivacaine deposited posterior to the quadratus lumborum muscle. 150mcg morphine will be added to the spinal anaesthetic.
  Arms: Intrathecal morphine as well as local anaesthetic in Blocks; Saline intrathecal as well as local anaesthetic in Blocks
Procedure: Intrathecal morphine as well as saline in Block — 150mcg morphine will be added to the spinal anaesthetic. 25 ml saline will be used on each side during a quadratus lumborum type 2 block.
  Arms: Intrathecal morphine as well as local anaesthetic in Blocks; Intrathecal morphine as well as saline in Block
Procedure: Saline intrathecal as well as saline in Blocks — 0.3 ml saline will be added to the spinal anaesthetic. 25 ml saline will be used on each side during a quadratus lumborum type 2 block.
  Arms: Saline intrathecal as well as local anaesthetic in Blocks; Saline intrathecal as well as saline in Blocks
Procedure: Saline intrathecal as well as local anaesthetic in Blocks — 0.3 ml saline will be added to the spinal anaesthetic. A Quadratus lumborum type 2 block will be performed under ultrasound with 25 ml 0.375% ropivacaine deposited posterior to the quadratus lumborum muscle.
  Arms: Intrathecal morphine as well as saline in Block; Saline intrathecal as well as saline in Blocks

SUMMARY:
The investigators are comparing post operative analgesia provided for caesarean section patients, with the quadratus lumborum type 2 block and intrathecal morphine.

DETAILED DESCRIPTION:
In Australia the rate of birth via caesarean section (CS) has significantly increased over the last twenty years. Improvements in the care of women undergoing CS are important locally, nationally and internationally. Compared to women birthing vaginally, women undergoing CS experience more adverse events and more pain. Effective pain relief following CS is important as it enables early ambulation, encourages maternal bonding, and promotes breastfeeding initiation and establishment. Traditional analgesic techniques following CS include opioid medications. Whist effective, the use of opioids are associated with frequent and significant side effects. Alternative analgesic agents are being explored in an attempt to improve the effectiveness of pain relief available to women and clinicians.

The quadratus lumborum block (QLB) block is an innovative regional analgesic technique. Its role as an effective analgesic agent in abdominal surgery is increasing. However, it has not been studied for pain relief in Australia after cesarean section.

In this study, the investigator aims to compare post-operative analgesia and side effects between the QLB blocks versus adding morphine the participant's spinal anaesthetic (ITM) during the elective C/S. Results from this study will provide information on the analgesic impact of this new and emerging therapy and assist in the development of a larger clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Anaesthetist trained in QLB and ITM techniques available
* American Society of Anaesthesiologists PS category client I or II
* 18 years of age or older
* Ability to read and understand English
* Uncomplicated pregnancy at term (>37 weeks completed gestation)
* Booked elective CS

Exclusion Criteria:

* Contraindications to spinal anaesthesia
* History of chronic opioid consumption / chronic pain conditions
* Known allergy to study drugs
* Weight more than 95kg or body mass index (BMI) more than 35 pre operative
* Placenta Previa / accreta
* Obstructive Sleep apnoea
* Severe asthma unable to tolerate Non steroidal anti inflammatory agents

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female patients undergoing elective cesarean sections
Enrollment: 0 (Actual)
Dates: Start 2019-01-01 (Estimated); Primary Completion 2019-11-01 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
24 hours total intravenous morphine usage via a PCA pump | 24 hours
  Post operative intravenous morphine use will be noted at 24 hours post cesarean section

SECONDARY OUTCOMES:
Patient's side effects within the 24 hours post operative period. | 24 hours
  Nausea, vomiting, itching, herpes reactivation, urinary retention and sedation will be noted.
Pain Scores within 24 hours post operative period. | 24 hours
  Using a VAS we will note both dynamic and static pain scores at 24 hours post operative

CONTACTS AND LOCATIONS:
Overall Officials: Willem Basson, FANZCA, Principal Investigator — Sunshine Coast University Hospital

IPD SHARING:
Plan to Share IPD: No